CLINICAL TRIAL: NCT05788913
Title: Randomized, Open-label, Single-dose, Crossover Study to Evaluate the Pharmacodynamics of an Unfractionated Heparin Compared to Heparin Sodium Injection, USP (Comparator) After Subcutaneous Administration in Healthy Subjects
Brief Title: Evaluation of the Pharmacodynamics of a Heparin With Its Biological Comparator, Subcutaneous Administration
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Blau Farmaceutica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CAEP 98.002.22
Record Dates: First submitted 2023-01-27; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Anticoagulant
MeSH Terms: interventions — Heparin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference Drug (Active Comparator): Healthy participants using intravenous Heparin Sodium Injection, USP (Fresenius Kabi) to assess the pharmacodynamic profile
  Interventions: Biological: Heparin
- Test Drug (Experimental): Healthy participants using intravenous Heparin Test to assess the pharmacodynamic profile
  Interventions: Biological: Heparin

INTERVENTIONS:
Biological: Heparin — subcutaneous Heparin

SUMMARY:
Experimental Drug: Porcine sodium heparin, injectable solution - 5,000 IU/ 0.25 mL; Blau Farmacêutica S/A.

Comparator Drug: Heparin Sodium Injection, USP, injectable solution - 5,000 IU/ 0.5 mL; Fresenius Kabi Lake Zurich.

Evaluate the equivalence in terms of pharmacodynamics of heparin sodium (test product) and Heparin Sodium Injection, USP (comparator product). The clinical trial will last approximately 08 weeks and the study population will consist of 68 healthy research participants, 34 women and 34 men

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent approved by a Research Ethics Committee (CEP) prior to any trial-related activities;
2. Healthy male or female participants between 18 and 55 years of age;
3. Be in good health or have no significant illness at the discretion of the responsible researcher/physician, in accordance with what is defined in this protocol and the assessments to which he/she is submitted during recruitment and selection, such as: clinical history, vital signs, anthropometric data, physical examination , ECG and laboratory tests;
4. Have a Body Mass Index (BMI) ≥ 18.5 and ≤ 29.9 Kg/m2, inclusive;
5. Present body weight between 60 and 100 Kg;
6. Agree to abstain from alcohol consumption for the duration of the study;
7. Present a negative result for the test for detecting alcohol in urine or saliva;
8. Test negative for the coronavirus (SARS-CoV-2);
9. Be able to understand the nature and purpose of the study, including risks and adverse events;
10. Act in accordance with the requirements of the entire trial, which is confirmed by signing the Free and Informed Consent Form (TCLE);
11. The drug can bring serious risks to the fetus, so the research participant, whether female or male, must agree to use a safe contraceptive method. Male participants must refrain from donating sperm from admission to final visit

Exclusion Criteria:

1. Present flu-like symptoms that, at the physician's discretion, are suspected of being infected by the coronavirus within 7 days prior to the period of hospitalization;
2. Having had direct and significant contact at medical discretion with people who tested positive for the coronavirus (SARS-CoV-2) test within 14 days prior to the hospitalization period;
3. Known to have a hypersensitivity reaction to the studied drug, pork foods or chemically related compounds;
4. Have used regular medication within 14 days prior to the hospitalization period;
5. Have used any medication within 7 days prior to the hospitalization period, except for contraceptives, cases in which, based on the half-life of the drug and/or active metabolites, complete elimination can be assumed or that, at the discretion of the responsible investigator/physician does not interfere in the pharmacokinetics or in the analytical stage of the study drug;
6. Having received any vaccine dose within 7 days prior to the hospitalization period;
7. Have received, within the three months prior to the study, treatment with any drug known to have well-defined toxic potential in large organs;
8. Have participated in any experimental study or ingested any experimental drug within the six months prior to the start of this study;
9. Have been hospitalized for any reason up to eight weeks before the start of the first treatment period of this study;
10. Have a history of liver, gastrointestinal or other conditions that may interfere with the absorption, distribution, metabolism or excretion of the drug;
11. Have a history of renal, respiratory, hematological, cardiological, neurological, neoplastic or psychiatric disease considered clinically significant at the physician's discretion;
12. Have a history of cardiac surgery (whatever), renal (renal exeresis or agenesis), gastrointestinal (partial or total removal of the esophagus, stomach, duodenum, jejunum, ileum, ascending colon, transverse colon, descending colon, sigmoid and rectum ) and surgery of the liver or pancreas;
13. Have any current symptom or disease, acute or chronic, being monitored or treated, significant at the discretion of the responsible researcher/physician;
14. Possess any active systemic or immunological disease or condition, including but not limited to the following general categories: cardiovascular/pulmonary, hepatic, renal or systemic infection or lactation;
15. Electrocardiographic findings not recommended at the physician's discretion for participation in the study;
16. Have the results of laboratory tests performed in the clinical evaluation of recruitment outside the values considered normal according to the reference values stipulated by the clinical analysis laboratory, unless they are considered not clinically significant by the researcher in charge/physician;
17. Have results of laboratory tests that, according to medical evaluation, affect the safety of the research participant;
18. Present clinically significant abnormalities on physical examination;
19. Have donated blood in the last 30 days;
20. Individuals taking aspirin or any other non-steroidal anti-inflammatory agent, with or without a doctor's prescription, within 10 days of treatment;
21. Clinically significant abnormality in vital signs or electrocardiogram (ECG), as judged by the investigator;
22. Known allergic or undesirable reactions following the use of unfractionated heparin;
23. Subjects who will undergo any surgical procedure within 14 days after the conclusion of the study;
24. Failure to show up for the coronavirus (SARS-CoV-2) test before admission;
25. Present a positive or inconclusive test for the coronavirus before admission;
26. Present a positive test for pregnancy during pre-hospitalization;
27. Present a positive result for the test for alcohol detection through urine or saliva;
28. Have a positive preliminary drug test with methamphetamine, opiate/morphine, marijuana/tetrahydrocannabinol, amphetamine, cocaine/benzoylecgonine and/or benzodiazepine;
29. Being a smoker or having quit smoking less than 6 months ago;
30. Have a history of illicit drug abuse;
31. Have an average alcohol intake of more than 3 alcoholic drinks in one day, or more than 7 alcoholic drinks per week, for women and more than 4 alcoholic drinks in one day, or more than 14 alcoholic drinks alcoholic beverages per week, for men;
32. Have consumed alcohol and/or drugs in the 48 hours prior to the period of hospitalization;
33. Having the habit of drinking more than five cups of coffee or tea a day;
34. Ingest food or drinks containing xanthines in the 48 hours prior to hospitalization;
35. Having done some intense physical exercise in the 48 hours prior to hospitalization;
36. Having unusual eating habits or with restrictions at the discretion of the responsible researcher/physician;
37. Be pregnant or breastfeeding, suspect pregnancy or wish to become pregnant while conducting the study;
38. Have donated or lost 450 mL or more of blood in the last three months;
39. Have donated or lost more than 1500 mL of blood in the last twelve months;
40. Show inability to stay awake or lying down for 1 hour or time required at the doctor's discretion;
41. Have any condition that prevents participation in the study at the discretion of the researcher in charge/physician;
42. Research participant who has participated in clinical trial protocols in the last 12 (twelve) months (CNS Resolution 251, of August 7, 1997, item III, subitem J).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Amax parameter pharmacodynamics for the anti-FXA marker | 12 hours of blood collection from the administration of the test drug and 12 hours of blood collection from the administration of the reference drug. The doses will be separated by a minimum interval of 14 days.
  Amax: Maximum response, understood as the highest concentration, detected in plasma after treatment.
  The conclusion by the average equivalence is achieved when the confidence intervals 90% of the ratio of geometric averages of experimental and comparator drugs are between 80% and 125%.
Evaluation of ASCE0-t parameter pharmacodynamics for the anti-FXA marker | 12 hours of blood collection from the administration of the test drug and 12 hours of blood collection from the administration of the reference drug. The doses will be separated by a minimum interval of 14 days.
  ASCE0-T: area under the effect-based effect curve versus time from zero to the last experimentally determined concentration;
  The conclusion by the average equivalence is achieved when the confidence intervals 90% of the ratio of geometric averages of experimental and comparator drugs are between 80% and 125%.
Evaluation of ASCE0-inf parameter pharmacodynamics for the anti-FXA marker | 12 hours of blood collection from the administration of the test drug and 12 hours of blood collection from the administration of the reference drug. The doses will be separated by a minimum interval of 14 days.
  ASCE0-inf: Area under the effect curve based on concentration versus time from zero to infinity experimentally determined.
  The conclusion by the average equivalence is achieved when the confidence intervals 90% of the ratio of geometric averages of experimental and comparator drugs are between 80% and 125%.
Evaluation of Amax parameter pharmacodynamics for the anti-FIIA marker | 12 hours of blood collection from the administration of the test drug and 12 hours of blood collection from the administration of the reference drug. The doses will be separated by a minimum interval of 14 days.
  Amax: Maximum response, understood as the highest concentration, detected in plasma after treatment.
  The conclusion by the average equivalence is achieved when the confidence intervals 90% of the ratio of geometric averages of experimental and comparator drugs are between 80% and 125%.
Evaluation of ASCE0-t parameter pharmacodynamics for the anti-FIIA marker | 12 hours of blood collection from the administration of the test drug and 12 hours of blood collection from the administration of the reference drug. The doses will be separated by a minimum interval of 14 days.
  ASCE0-T: area under the effect-based effect curve versus time from zero to the last experimentally determined concentration;
  The conclusion by the average equivalence is achieved when the confidence intervals 90% of the ratio of geometric averages of experimental and comparator drugs are between 80% and 125%.

SECONDARY OUTCOMES:
Sequence effects of pharmacodynamic parameters for the Anti-FXa marker - Analysis of variance (ANOVA) | 12 hours of blood collection from the administration of the test drug and 12 hours of blood collection from the administration of the reference drug. The doses will be separated by a minimum interval of 14 days.
  Amax and ASCEo-t and ASCEo-inf parameters will be analyzed by analyzing ANOVA variance to evaluate the sequence effects of the anti-fii marker
Sequence effects of pharmacodynamic parameters for the Anti-FIIa marker - Analysis of variance (ANOVA) | 12 hours of blood collection from the administration of the test drug and 12 hours of blood collection from the administration of the reference drug. The doses will be separated by a minimum interval of 14 days.
  Amax and ASCEo-t parameters will be analyzed by analyzing ANOVA variance to evaluate the sequence effects of the anti-fii marker
Ratio of Anti-FXa/Anti-FIIa activity based on the pharmacodynamic parameter ASCE0-t | 12 hours of blood collection from the administration of the test drug and 12 hours of blood collection from the administration of the reference drug. The doses will be separated by a minimum interval of 14 days.
  The ratio for anti-FXa/anti-FIIa activity of the ASCE0-t parameter will be evaluated. , the evaluation will be performed by comparing the interval of 90% of the ratio with the equivalence criterion 80% - 125%.
Occurrence of adverse events and serious eventsevents | 2 months
  Adverse events will be monitored for two months and reported in the final report.
  * Total of adverse events;
  * Total number of research participants who had adverse events;
  * Number of adverse events per period;
  * Number of adverse events due to causality;
  * Number of adverse events by type of medicine (formulation);
  * Number of adverse EA intensity events.
Evaluation of Amax parameter pharmacodynamics for the tissue factor pathway inhibitor (TFPI) activity | 12 hours of blood collection from the administration of the test drug and 12 hours of blood collection from the administration of the reference drug. The doses will be separated by a minimum interval of 14 days.
  TFPI serum concentrations will be quantified by ELISA method.
  will be evaluated by comparing the 90% interval for the ratios with the acceptance criteria 80% - 125%.
Evaluation of ASCEo-t parameter pharmacodynamics for the tissue factor pathway inhibitor (TFPI) activity | 12 hours of blood collection from the administration of the test drug and 12 hours of blood collection from the administration of the reference drug. The doses will be separated by a minimum interval of 14 days.
  TFPI serum concentrations will be quantified by ELISA method.
  will be evaluated by comparing the 90% interval for the ratios with the acceptance criteria 80% - 125%.
Evaluation of ASCEo-inf parameter pharmacodynamics for the tissue factor pathway inhibitor (TFPI) activity | 12 hours of blood collection from the administration of the test drug and 12 hours of blood collection from the administration of the reference drug. The doses will be separated by a minimum interval of 14 days.
  TFPI serum concentrations will be quantified by ELISA method.
  will be evaluated by comparing the 90% interval for the ratios with the acceptance criteria 80% - 125%.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Research, Study Director — Blau Farmaceutica S.A.